CLINICAL TRIAL: NCT04730804
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study of Subcutaneous ALXN1830 in Healthy Participants
Brief Title: A Study of ALXN1830 in Healthy Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to terminate program
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ALXN1830-HV-108
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: ALXN1830; Autoimmune Disease; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Autoimmune Diseases | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Cohort 1: ALXN1830 Single Dose 1/Placebo (Experimental): Participants will receive a single SC dose of ALXN1830 or placebo.
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 2: ALXN1830 Single Dose 2/Placebo (Experimental): Participants will receive a single SC dose of ALXN1830 or placebo.
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 3: ALXN1830 Multiple Dose 1/Placebo (Experimental): Participants will receive multiple SC doses of ALXN1830 or placebo.
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 4: ALXN1830 Multiple Dose 2/Placebo (Experimental): Participants will receive multiple SC doses of ALXN1830 or placebo.
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 5: ALXN1830 Multiple Dose 3/Placebo (Experimental): Participants will receive multiple SC doses of ALXN1830 or placebo.
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 6: ALXN1830 /Placebo in Japanese Population (Experimental): Japanese participants will receive multiple SC doses of ALXN1830 (HTD) or placebo.
  Interventions: Drug: ALXN1830; Drug: Placebo

INTERVENTIONS:
Drug: ALXN1830 — ALXN1830 will be administered as SC infusion(s).
Drug: Placebo — Placebo will be administered as SC infusion(s).
  Other Names: Normal Saline

SUMMARY:
This trial will study the effects of single and multiple doses of ALXN1830 in healthy adult participants.

DETAILED DESCRIPTION:
This is a Phase 1 study in healthy adult participants. The study will consist of 2 single ascending dose (Cohorts 1 and 2) and 4 multiple ascending dose cohorts (Cohorts 3 to 6). Participants will be randomly assigned to each of the 6 cohorts to receive either single or multiple doses of ALXN1830 subcutaneous (SC) or single or multiple doses of placebo SC. Cohort 6 will enroll only healthy participants of Japanese descent who will be dosed according to the highest tolerated dose (HTD) established in the non-Japanese cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Satisfactory medical assessment.
* Participants must have had vaccination against pneumococcus (Pneumovax 23 [PPSV23]) at least 28 days, and maximally 4 years prior to Day 1.
* Participants must have had seasonal influenza vaccination for the current season at least 28 days prior to Day 1.
* Body weight within 60 to 90 kilograms (kg), inclusive, and body mass index within 18 to 30 kg/meter squared, inclusive.
* Must be willing to follow protocol-specified contraception guidance during the study and for 3 months after last dose of study drug.

Exclusion Criteria:

* Current/recurrent diseases or relevant medical history.
* Known exposure to investigational or marketed therapeutic proteins, such as monoclonal antibodies, fusion proteins, bispecific molecules, or antibody drug conjugates, within 60 days or 5 half-lives (whichever is longer) prior to dosing.
* Participants who have prior exposure to ALXN1830.
* Current enrollment or past participation within the last 90 days before signing of consent in this or any other interventional clinical study.
* Participants with hepatitis B or C, or human immunodeficiency virus.
* Participants who are either immunocompromised or have one of the following underlying medical conditions: anatomic or functional asplenia (including sickle cell disease); primary antibody deficiencies.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Clinical Trial Site, Auckland
  - Research Site, Grafton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1830-HV-108&attachmentIdentifier=06168a24-b6da-4060-9d5a-c64a34424d7d&fileName=ALXN1830-HV-108_CSR_Synopsis_Final_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 34 participants (25 ALXN1830 treated and 9 placebo-treated) were enrolled and randomized in a 6:2 ratio in 5 cohorts. Healthy, Japanese participants were planned to be dosed in Cohort 6 according to the highest tolerated dose (HTD) established in the non-Japanese cohorts. This cohort was not achieved due to early termination of the study.
Groups:
- Cohort 1: ALXN1830 Single Medium Dose: Participants received a single subcutaneous (SC) medium dose of ALXN1830.
- Cohort 2: ALXN1830 Single Hign Dose: Participants received a single SC high dose of ALXN1830.
- Cohort 3: ALXN1830 Multiple Low Dose: Participants received multiple SC low doses of ALXN1830 once weekly (QW).
- Cohort 4: ALXN1830 Multiple Medium Dose: Participants received multiple SC medium doses of ALXN1830 QW.
- Cohort 5: ALXN1830 Multiple High Dose: Participants received multiple SC high doses of ALXN1830 QW.
- Placebo: Participants received placebo matched to ALXN1830.
Period: Overall Study
Arm/Group | Cohort 1: ALXN1830 Single Medium Dose | Cohort 2: ALXN1830 Single Hign Dose | Cohort 3: ALXN1830 Multiple Low Dose | Cohort 4: ALXN1830 Multiple Medium Dose | Cohort 5: ALXN1830 Multiple High Dose | Placebo
Started | 6 | 1 | 6 | 6 | 6 | 9
Received at Least 1 Dose of Study Drug | 6 | 1 | 6 | 6 | 6 | 9
Completed | 6 | 1 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who received at least 1 dose of study drug.
Groups:
- Cohort 1: ALXN1830 Single Medium Dose: Participants received a single SC medium dose of ALXN1830.
- Cohort 2: ALXN1830 Single High Dose: Participants received a single SC high dose of ALXN1830.
- Cohort 3: ALXN1830 Multiple Low Dose: Participants received multiple SC low doses of ALXN1830 QW.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ALXN1830 Single Medium Dose | Cohort 2: ALXN1830 Single High Dose | Cohort 3: ALXN1830 Multiple Low Dose | Cohort 4: ALXN1830 Multiple Medium Dose | Cohort 5: ALXN1830 Multiple High Dose | Placebo | Total
Number analyzed (Participants) | 6 | 1 | 6 | 6 | 6 | 9 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 1 | 6 | 6 | 6 | 9 | 34
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 2 | 3 | 5 | 17
  Male | 3 | 0 | 3 | 4 | 3 | 4 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 5 | 0 | 4 | 3 | 3 | 4 | 19
  Race: Asian Indian | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Race: Chinese | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Race: Other Asian | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Race: Samoan | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Race: Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Race: Other | 1 | 1 | 1 | 2 | 1 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not of Hispanic, Latino/a, or Spanish origin | 4 | 0 | 4 | 4 | 6 | 5 | 23
  Ethnicity: Another Hispanic, Latino/a, or Spanish origin | 0 | 0 | 0 | 1 | 0 | 2 | 3
  Ethnicity: Not Reported | 1 | 1 | 1 | 1 | 0 | 1 | 5
  Ethnicity: Unknown | 1 | 0 | 1 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant administered the study drug and which did not necessarily have a causal relationship with this treatment. A TEAE was defined as an AE with a start date or time on or after the first dose of the study intervention. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Day 1 (postdose) through follow-up (up to approximately 141 days)
Population: The Safety Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1830 Single Medium Dose | Cohort 2: ALXN1830 Single High Dose | Cohort 3: ALXN1830 Multiple Low Dose | Cohort 4: ALXN1830 Multiple Medium Dose | Cohort 5: ALXN1830 Multiple High Dose | Placebo
Number analyzed (Participants) | 6 | 1 | 6 | 6 | 6 | 9
Participants | 6 | 1 | 6 | 6 | 5 | 7

2. Secondary Outcome: Single-Dose Cohorts: Area Under the Serum Concentration-time Curve From Time 0 (Dosing) To Time Infinity (AUC0-inf) of ALXN1830
Description: Serum total drug concentrations were measured using a validated liquid chromatography/mass spectrometry (LC/MS) assay.
Time Frame: Day 1 (predose) up to Day 64 (postdose)
Population: The Pharmacokinetic Set included all participants who received at least 1 dose of study drug (only active) and had at least 1 postdose serum ALXN1830 concentration measured. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*milligram (mg)/liter (L)
Arm/Group | Cohort 1: ALXN1830 Single Medium Dose | Cohort 2: ALXN1830 Single High Dose
Number analyzed (Participants) | 1 | 1
hours*milligram (mg)/liter (L) | 360.940 | 291.930

3. Secondary Outcome: Multiple-Dose Cohorts: AUC0-inf of ALXN1830 at Day 1
Description: Serum total drug concentrations were measured using a validated LC/MS assay.
Time Frame: Day 1 (predose up to 12 hours postdose)
Population: The Pharmacokinetic Set included all participants who received at least 1 dose of study drug (only active) and had at least 1 postdose serum ALXN1830 concentration measured. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. Per prespecified analysis, only participants in Cohort 5 were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*mg/L
Arm/Group | Cohort 3: ALXN1830 Multiple Low Dose | Cohort 4: ALXN1830 Multiple Medium Dose | Cohort 5: ALXN1830 Multiple High Dose
Number analyzed (Participants) | 0 | 0 | 4
hours*mg/L |  |  | 340.085 (162.0531)

4. Secondary Outcome: Multiple-Dose Cohorts: AUC0-inf of ALXN1830 at Day 22
Description: Serum total drug concentrations were measured using a validated LC/MS assay.
Time Frame: Day 22 (predose up to 12 hours postdose)
Population: The Pharmacokinetic Set included all participants who received at least 1 dose of study drug (only active) and had at least 1 postdose serum ALXN1830 concentration measured. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. Per prespecified analysis, only participants in Cohort 4 were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*mg/L
Arm/Group | Cohort 3: ALXN1830 Multiple Low Dose | Cohort 4: ALXN1830 Multiple Medium Dose | Cohort 5: ALXN1830 Multiple High Dose
Number analyzed (Participants) | 0 | 3 | 0
hours*mg/L |  | 333.787 (143.7390) |

5. Secondary Outcome: Multiple-Dose Cohorts: AUC0-inf of ALXN1830 at Day 78
Description: Serum total drug concentrations were measured using a validated LC/MS assay.
Time Frame: Day 78 (predose up to 12 hours postdose)
Population: The Pharmacokinetic Set included all participants who received at least 1 dose of study drug (only active) and had at least 1 postdose serum ALXN1830 concentration measured. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint. Per prespecified analysis, only participants in Cohort 3 were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*mg/L
Arm/Group | Cohort 3: ALXN1830 Multiple Low Dose | Cohort 4: ALXN1830 Multiple Medium Dose | Cohort 5: ALXN1830 Multiple High Dose
Number analyzed (Participants) | 1 | 0 | 0
hours*mg/L | 847.380 |  |

6. Secondary Outcome: Change From Baseline in Serum Immunoglobulin G (IgG) at Early Termination Visit (up to Day 141)
Description: Serum concentration of IgG was measured using validated nephelometric assays.
Time Frame: Baseline, early termination visit (up to Day 141)
Population: The Pharmacodynamic Set included all participants who received at least 1 dose of study drug (active and placebo) who had evaluable serum Immunoglobulin data (IgG, IgG subtypes, Ig subtypes, and circulating immune complexes [CIC]) or neonatal crystallizable fragment receptor (FcRn) data.
Measure: Mean (Standard Deviation); unit: grams (g)/L
Arm/Group | Cohort 1: ALXN1830 Single Medium Dose | Cohort 2: ALXN1830 Single High Dose | Cohort 3: ALXN1830 Multiple Low Dose | Cohort 4: ALXN1830 Multiple Medium Dose | Cohort 5: ALXN1830 Multiple High Dose | Placebo
Number analyzed (Participants) | 6 | 1 | 6 | 6 | 6 | 9
grams (g)/L | -0.60 (1.037) | -1.00 | -0.22 (1.504) | -0.70 (0.899) | 0.10 (0.555) | -0.17 (1.122)

7. Secondary Outcome: Percent FcRN Receptor Occupancy at Day 120
Time Frame: Day 120
Population: The Pharmacodynamic Set included all participants who received at least 1 dose of study drug (active and placebo) who had evaluable serum Immunoglobulin data (IgG, IgG subtypes, Ig subtypes, and CIC) or FcRn data. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of receptor occupied
Arm/Group | Cohort 1: ALXN1830 Single Medium Dose | Cohort 2: ALXN1830 Single High Dose | Cohort 3: ALXN1830 Multiple Low Dose | Cohort 4: ALXN1830 Multiple Medium Dose | Cohort 5: ALXN1830 Multiple High Dose | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 0 | 0 | 1
percentage of receptor occupied |  |  | 12.07 (92.0) |  |  | 6.40

8. Secondary Outcome: Number of Participants With Antidrug Antibodies (ADA) and Neutralizing Antibodies (NAb) to ALXN1830
Time Frame: Day 1 (postdose) through follow-up (up to approximately 141 days)
Population: The Immunogenicity Set included all participants who had a predose (baseline) and at least 1 postdose ADA sample collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1830 Single Medium Dose | Cohort 2: ALXN1830 Single High Dose | Cohort 3: ALXN1830 Multiple Low Dose | Cohort 4: ALXN1830 Multiple Medium Dose | Cohort 5: ALXN1830 Multiple High Dose | Placebo
Number analyzed (Participants) | 6 | 1 | 6 | 6 | 6 | 9
Participants
  ADA positive | 6 | 1 | 6 | 6 | 5 | 6
  NAb | 4 | 0 | 6 | 4 | 2 | 2

ADVERSE EVENTS:
Time Frame: Day 1 (postdose) through follow-up (up to approximately 141 days)
Description: The Safety Set included all participants who received at least 1 dose of study drug.
Arm/Group | Cohort 1: ALXN1830 Single Medium Dose | Cohort 2: ALXN1830 Single High Dose | Cohort 3: ALXN1830 Multiple Low Dose | Cohort 4: ALXN1830 Multiple Medium Dose | Cohort 5: ALXN1830 Multiple High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/1 | 0/6 | 0/6 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/1 | 0/6 | 0/6 | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 6/6 | 1/1 | 6/6 | 6/6 | 5/6 | 7/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ALXN1830 Single Medium Dose (N=6) | Cohort 2: ALXN1830 Single High Dose (N=1) | Cohort 3: ALXN1830 Multiple Low Dose (N=6) | Cohort 4: ALXN1830 Multiple Medium Dose (N=6) | Cohort 5: ALXN1830 Multiple High Dose (N=6) | Placebo (N=9)
Injection site erythema (General disorders) | 2 | 1 | 5 | 6 | 2 | 1
Injection site pain (General disorders) | 0 | 1 | 3 | 3 | 2 | 0
Injection site swelling (General disorders) | 4 | 1 | 2 | 2 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 2 | 2 | 1 | 0
Injection site induration (General disorders) | 0 | 0 | 1 | 2 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 3 | 1 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Catheter site vesicles (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site paraesthesia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site urticaria (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mass (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Medical device site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 3 | 4 | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 3 | 0 | 1
Acarodermatitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gonorrhoea (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 3 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT04730804/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT04730804/SAP_001.pdf